CLINICAL TRIAL: NCT03834831
Title: Impact of Coenzyme Q10 and Selenium on Seminal Fluid Parameters and Antioxidant Status in Men With Idiopathic Infertility
Brief Title: Impact of Coenzyme Q10 and Selenium on Seminal Fluid and Semen Antioxidant Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sumer (Other)
Responsible Party: Principal Investigator, Dr. Ahmed T Alahmar, Principal Investigator, University of Sumer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC/2018/8866
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Male Infertility
Keywords: Male infertility; Coenzyme Q10; Selenium; Antioxidants
MeSH Terms: conditions — Infertility, Male | interventions — coenzyme Q10; Selenium

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coenzyme Q10 (Active Comparator): Coenzyme Q10 200mg/day for 3 months
  Interventions: Dietary Supplement: Coenzyme Q10
- Selenium (Active Comparator): Selenium mcg/day for 3 months
  Interventions: Dietary Supplement: Selenium

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — Coenzyme Q10
  Arms: Coenzyme Q10
Dietary Supplement: Selenium — Selenium
  Arms: Selenium

SUMMARY:
The study was conducted to assess the impact of coenzyme Q10 and selenium on seminal fluid parameters and antioxidant status in infertile men.

DETAILED DESCRIPTION:
The aim of this study was to assess the impact of coenzyme Q10 and selenium on seminal fluid parameters and antioxidant status in infertile men with idiopathic oligoasthenoteratospermia.

ELIGIBILITY:
Inclusion Criteria:

* History of infertility of at least 12 months despite regular unprotected intercourse.
* Oligoasthenoteratospermia was diagnosed by semen analysis showing abnormal sperm concentration (<15 million/ml), progressive motility (<32%), total motility (<40%) and morphology (<30% WHO criteria) as defined by WHO manual for semen analysis 2010

Exclusion Criteria:

* Azoospermia,
* Varicocele,
* Genital tract infection,
* Cryptorchidism,
* Testicular trauma or scrotal surgery,
* Endocrine disorder,
* Systemic illness,
* Smoking
* The presence of female factor

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male infertility
Enrollment: 70 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Semen volume (WHO 2010 guidelines) | 3 months
  Semen volume in ml
Sperm concentration in semen (WHO 2010 guidelines) | 3 months
  Sperm concentration in million/ml
Sperm motility in semen (WHO 2010 guidelines) | 3 months
  Sperm motility (%)
Sperm morphology in semen (WHO 2010 guidelines) | 3 months
  Normal sperm morphology (%)
Seminal plasma TAC (Colorimetric assays) | 3 months
  Seminal plasma total antioxidant capacity in mmol/ml
Seminal plasma CAT (Colorimetric assays) | 3 months
  Seminal plasma catalase in U/ml
Seminal plasma SOD (Colorimetric assays) | 3 months
  Superoxide dismutase in U/ml

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed T Alahmar, Principal Investigator — University of Sumer, Iraq
Locations (1):
- Fertility Unit, Babyl, Hillah, Iraq

IPD SHARING:
Plan to Share IPD: No
Patients data are anonymous and in hold with the principal investigator

REFERENCES:
- [Background] Alshahrani S, Aldossari K, Al-Zahrani J, Gabr AH, Henkel R, Ahmad G. Interpretation of semen analysis using WHO 1999 and WHO 2010 reference values: Abnormal becoming normal. Andrologia. 2018 Mar;50(2). doi: 10.1111/and.12838. Epub 2017 Aug 3. PMID 28771785
- [Background] Alahmar AT. The effects of oral antioxidants on the semen of men with idiopathic oligoasthenoteratozoospermia. Clin Exp Reprod Med. 2018 Jun;45(2):57-66. doi: 10.5653/cerm.2018.45.2.57. Epub 2018 Jun 29. PMID 29984205